CLINICAL TRIAL: NCT00844922
Title: Double-blind, Placebo-controlled Trial Investigating the Safety of Re-exposure to 900 mg of Org 34517, Used as Adjunctive Therapy in Subjects With Psychotic Major Depression (Major Depressive Episode, Severe, With Psychotic Features), Who Participated in Trial 28130
Brief Title: Safety of Org 34517 900 mg in Patients Who Received Org 34517 in a Previous Trial (Study 28133/P05842)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05842; EudraCT #: 2004-002156-34;; P05842
Record Dates: First submitted 2009-02-11; First posted 2009-02-16 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Depressive Disorders; Psychotic Disorders; Depression
MeSH Terms: conditions — Depressive Disorder; Psychotic Disorders; Depression | interventions — Org 34517

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Org 34517 (Experimental): Org 34517 titrated to 900 mg daily for 2 weeks
  Interventions: Drug: SCH 900636
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCH 900636 — Org 34517 300 mg on Day 1, 600 mg on Day 2, then 900 mg daily starting from Day 3. Subjects in this arm were also to continue the "usual treatment" for psychotic major depression.
  Other Names: Org 34517
  Arms: Org 34517
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Patients who participated in the previous trial 28130, who were eligible, were entered into this trial. Patients who were randomized to placebo in the previous trial 28130 continued on placebo while patients who were randomized to Org 34517 (SCH 900636), regardless of dose, were titrated to 900 mg Org 34517. Patients in this trial took their study medication for 2 weeks in order to study the safety and tolerability of Org 34517.

ELIGIBILITY:
Inclusion Criteria:

* have attended Screening, Baseline, Visit Day 15, Day 29 and Day 43 of previous trial 28130;
* have a CGI of Severity score of 3 or greater at Day 43 of previous trial 28130 and at Day 1 of current trial 28133, or a lower score when the investigator is of the opinion that further resolution of symptoms is warranted;
* be on a stable dose of 'usual treatment', which must consist of an antidepressant, an antipsychotic, a mood stabilizer or any combination of these 3 drug classes.

Exclusion Criteria:

* had experienced any of the following significant safety outcomes in previous trial 28130:

  * severe breakthrough bleeding;
  * diagnosis of prostatitis;
  * abnormal level of testosterone at Day 15 of previous trial 28130;
  * any adverse event deemed relevant for exclusion in trial 28133 by the investigator.
* had an abnormal PSA test at Day -7 of previous trial 28133
* were at significant risk of committing suicide, as indicated by a score greater than 9 on the revised ISST at Day -7 or Day 1;
* were currently treated with carbamazepine or valproate, midazolam, or clozapine;
* had been treated with electroconvulsive therapy (ECT) in the current episode;
* were currently treated with more than one antidepressant, antipsychotic, or mood stabilizer;
* had 'usual treatment' started or discontinued in the 2 weeks before Day 1;
* had a 'usual treatment' dose change within one week prior to Day 1;
* had any clinically unstable or uncontrollable renal, hepatic, respiratory, hematological, cardiovascular or cerebrovascular disease that would put the patient at risk of safety or bias assessment of efficacy;
* had known hypersensitivity reactions to glucocorticoid antagonists;
* had any clinically significant abnormal laboratory data (e.g. aspartate amino transferase (ASAT) and/or alanine amino transferase (ALAT) values > 2x normal range upper limit) or ECG results, or a clinically significant abnormal outcome at the physical examination at Day -7;
* had a confirmed positive result on the drug screening test for any illicit drug, except cannabis, at Day -7;
* had any untreated or uncompensated clinically significant endocrine disorder;
* were using hormone replacement therapy at Day -7;
* required concomitant treatment with corticosteroids (topical use was allowed);
* women of childbearing potential without adequate contraception
* women with a positive pregnancy test at Day -7 or 1, or are breast feeding mothers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability measures (vital signs, AEs) | 4 weeks

SECONDARY OUTCOMES:
17-item Hamilton Rating Scale for Depression (HAMD) total score | 4 weeks
proportion of BPRS 30% responders; proportion of subjects with sustained BPRS 30% response | 4 weeks
proportion of HAMD 50% responders; proportion of subjects with sustained HAMD 50% response | 4 weeks
clinical global impression (CGI) | 4 weeks
PANNS total score | 4 weeks
PANSS positive scale score, PANSS negative scale score, PANSS general psychopathology score | 4 weeks